CLINICAL TRIAL: NCT06303440
Title: Effects of Virtual Reality Versus Motor Imagery on Balance, Gross Motor Function and Activities of Daily Living in Children With Cerebral Palsy.
Brief Title: Effects of Virtual Reality Versus Motor Imagery in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0288
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; Motor control; activities of daily living; randomized controlled trial
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as assessor of the study would be kept blind of the treatment groups to which patient will be allocated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Routine Physical Therapy+ Balance Training) (Other): The children will be provided with Routine Physical Therapy and Balance Training.
  Balance exercises will be provided for 15 minutes and 30 minutes of Routine physical therapy will be as strengthening and stretching exercises.
  Interventions: Other: Routine Physical Therapy+ Balance Training
- Group B (Virtual Reality + Routine Physical Therapy) (Experimental): The VR system consisted of a wall-mounted display, a Nintendo Wii box, a Wii remote, and a Wii Fit board. The participants will be instructed to stand on Wii Fit board while interacting with the VR system and playing the selected games and routine physical therapy of 30 minutes will be provided.
  Interventions: Other: Virtual Reality+ Routine Physical Therapy
- Group C (Motor Imagery+ Routine Physical Therapy) (Experimental): During the presentation of a video clip, patients will watch the video and afterwards try to do movement as same as shown in video
  Interventions: Other: Motor Imagery+ Routine Physical Therapy

INTERVENTIONS:
Other: Routine Physical Therapy+ Balance Training — Each session will be begun with routine PT treatment and lasted for 45 minutes in total. To start, the participants will be asked to do warm-up exercises, sitting comfortably on a chair with their backs and feet well supported, the participants will be instructed to breathe in and out. Warm-up exercises will be carried out for 5 minutes. Stretching exercises will be performed for 15 minutes per session, and stretches were held for 30 seconds with four repetitions of each of the following areas, shoulder flexors, elbow and wrist flexors, hip flexors, hip adductors, knee flexors, and calf, 10 seconds of rest period will be added after stretching of one muscle group. Participants will have a 15 minutes session of exercises neck holding on form roller for 1 minute with two repetitions, astride-sitting on foam roller for 2 minutes with four repetitions, weight on both hands on gym ball for 1 minute with two repetitions and hip adductors strengthening for 1 minute with three repetitions.
  Arms: Group A (Routine Physical Therapy+ Balance Training)
Other: Virtual Reality+ Routine Physical Therapy — The exercises will be selected, and the difficulty level will be gradually increased according to participant's performance. Starting from the penguin slide, they will progress to table tilt. Initially, each game will be played for 2 minutes per session. With the progression of performance, 4 minutes of table tilt will be added. While playing this game, a typical mobility pattern will be initiated, and balance will be improved. In the same week, the subjects performed single-leg extensions for 1 minutes. In the following weeks, Balance Bubble, Advanced step, and Basic Run will be added to the plan. The participants will perform these activities for 7 minutes per session. Treatment sessions then progressed to motor function games, including bowling, tennis, kicking, and boxing (least challenging to most challenging), with most treatment sessions ending with boxing will be provided for 7 minutes and routine physical therapy for 30 minutes as explained in control group.
  Arms: Group B (Virtual Reality + Routine Physical Therapy)
Other: Motor Imagery+ Routine Physical Therapy — The 15 minutes of Motor Imagery session will be provided to participants. It's a three step process that will be used to incorporate the technique.
  Step I, The self-recorded videos of the principal researcher performing a normal movements will be shown to participant.
  Step II, The participants will be asked to imagine movement with eyes closed, and breathe deeply.
  Step III The participants will be asked to perform the movement you watched in video and routine physical therapy of 30 minutes will be provided.
  During the presentation of a video clip, patients will watch the video and afterwards try to do movement as same as shown in video.
  Arms: Group C (Motor Imagery+ Routine Physical Therapy)

SUMMARY:
Cerebral palsy is a neurodevelopmental disorder caused by brain injury that appears in infancy, children have mostly issues of gross motor functions, and activities of daily living. Virtual Reality is an innovative technique for the improvement of balance and motor function in most of the neurological conditions. Motor Imagery is an ability to engage in the mental representation of a task consciously without generating a voluntary movement. The aim of this study is to determine the comparative effects of Virtual Reality and Motor Imagery on balance, gross motor function and activities of daily living in children with cerebral palsy.

DETAILED DESCRIPTION:
This randomized controlled trial will be conducted at Rising Sun Institute. The sample size calculated for this trial will be 75. The participants will be randomly allocated using online randomization tool into three groups; Group A will receive routine physical therapy (PT) for 30 minutes with additional selected exercises for 15 minutes, Group B will receive VR training for 15 minutes with routine PT for 30 minutes, and Group C will receive MI for 15 minutes and routine PT for 30 minutes. Each participant will receive treatment for three days on alternative days per week for 12 weeks. Gross Motor Function Scale (GMFCS) will be used for balance, Bruininks-Oseretsky Test of motor function Proficiency-2 (BOT-2 ) for motor function, and WeeFIM scale for ADLs at baseline, 8th week, 12th week, and at 16th week after discontinuation of treatment.

ELIGIBILITY:
Inclusion Criteria:

Children of 7-12 years of both genders, Children with Mini Mental Scale score >24.

Children with Gross motor function classification system (GMFCS) level I and II and able to follow and accept verbal instruction.

Exclusion Criteria: History of any Visual and Hearing Impairments, Virtual game phobia.

History of nerve, muscle, bone and joint diseases that seriously affect the movement function of the limbs and Children with history of severe cardiopulmonary disease, History of epilepsy, History of Fixed deformity of Lower limb. History of orthopaedic surgery and botulinum toxin injection.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Classification System | 12 weeks
  Gross Motor Function Classification System will be used to measure balance
Bruininks-Oseretsky Test of motor function Proficiency-2 | 12 Weeks
  It will be measured with Bruininks-Oseretsky Test of motor function Proficiency-2 for motor function.
Functional Independence Measure for Children | 12 Weeks
  Functional Independence Measure for Children scale will be used to determine the Activities of Daily Living improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, PhD-PT, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu J, Loprinzi PD, Ren Z. The Rehabilitative Effects of Virtual Reality Games on Balance Performance among Children with Cerebral Palsy: A Meta-Analysis of Randomized Controlled Trials. Int J Environ Res Public Health. 2019 Oct 28;16(21):4161. doi: 10.3390/ijerph16214161. PMID 31661938
- [Background] Nashner LM, Shumway-Cook A, Marin O. Stance posture control in select groups of children with cerebral palsy: deficits in sensory organization and muscular coordination. Exp Brain Res. 1983;49(3):393-409. doi: 10.1007/BF00238781. PMID 6641837
- [Background] Chen CL, Shen IH, Chen CY, Wu CY, Liu WY, Chung CY. Validity, responsiveness, minimal detectable change, and minimal clinically important change of Pediatric Balance Scale in children with cerebral palsy. Res Dev Disabil. 2013 Mar;34(3):916-22. doi: 10.1016/j.ridd.2012.11.006. Epub 2013 Jan 3. PMID 23291508
- [Background] Ortega-Martinez A, Palomo-Carrion R, Varela-Ferro C, Bagur-Calafat MC. Feasibility of a Home-Based Mirror Therapy Program in Children with Unilateral Spastic Cerebral Palsy. Healthcare (Basel). 2023 Jun 19;11(12):1797. doi: 10.3390/healthcare11121797. PMID 37372915
- [Background] Brien M, Sveistrup H. An intensive virtual reality program improves functional balance and mobility of adolescents with cerebral palsy. Pediatr Phys Ther. 2011 Fall;23(3):258-66. doi: 10.1097/PEP.0b013e318227ca0f. PMID 21829120
- [Background] Kashif M, Ahmad A, Bandpei MAM, Gilani SA, Hanif A, Iram H. Combined effects of virtual reality techniques and motor imagery on balance, motor function and activities of daily living in patients with Parkinson's disease: a randomized controlled trial. BMC Geriatr. 2022 Apr 30;22(1):381. doi: 10.1186/s12877-022-03035-1. PMID 35488213
- [Background] Saleem GT. Defining and measuring motor imagery in children: mini review. Front Psychol. 2023 Aug 16;14:1227215. doi: 10.3389/fpsyg.2023.1227215. eCollection 2023. PMID 37655192
- [Background] Collet C, Guillot A, Lebon F, MacIntyre T, Moran A. Measuring motor imagery using psychometric, behavioral, and psychophysiological tools. Exerc Sport Sci Rev. 2011 Apr;39(2):85-92. doi: 10.1097/JES.0b013e31820ac5e0. PMID 21206282
- [Background] Steenbergen B, Craje C, Nilsen DM, Gordon AM. Motor imagery training in hemiplegic cerebral palsy: a potentially useful therapeutic tool for rehabilitation. Dev Med Child Neurol. 2009 Sep;51(9):690-6. doi: 10.1111/j.1469-8749.2009.03371.x. PMID 19709140
- [Background] Steenbergen B, Jongbloed-Pereboom M, Spruijt S, Gordon AM. Impaired motor planning and motor imagery in children with unilateral spastic cerebral palsy: challenges for the future of pediatric rehabilitation. Dev Med Child Neurol. 2013 Nov;55 Suppl 4:43-6. doi: 10.1111/dmcn.12306. PMID 24237279
- [Background] Souto DO, Cruz TKF, Fontes PLB, Haase VG. Motor imagery in children with unilateral cerebral palsy: a case-control study. Dev Med Child Neurol. 2020 Dec;62(12):1396-1405. doi: 10.1111/dmcn.14672. Epub 2020 Sep 29. PMID 32996138